CLINICAL TRIAL: NCT07221019
Title: Single-Shot Exparel Versus Catheters for Lower Extremity Orthopedic Trauma Patients
Brief Title: Single Shot Exparel vs Catheters in Lower Extremity Trauma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCR256547
Record Dates: First submitted 2025-10-23; First posted 2025-10-27 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Fracture Dislocation of Ankle Joint; Fracture Leg; Fracture Femur; Fracture Lower Leg; Fracture
MeSH Terms: conditions — Femoral Fractures; Fractures, Bone | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel + Bupivacaine (Experimental)
  Interventions: Drug: Exparel + Bupivacaine
- Bupivacaine (Active Comparator)
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Patients will receive the ERAS standard of care which includes gabapentin, Tylenol, and Toradol or Celebrex preoperatively as well as 20 cc of 0.25% bupivacaine with 10 cc of Exparel injected in the adductor space followed by 30 cc of 0.25% bupivacaine with 10 cc of Exparel in the sciatic nerve block. Injections will be completed by an anesthesia provider using astandard aseptic technique with ultrasound guidance. A 22 gauge 5-10cm needle is inserted with direct visualization under ultrasound and 2-5 cc aliquots are injected with aspiration repeated to ensure no vascular injury or injection until a total of 30 cc is injected into the adductor space and 40 cc is injected into the area surrounding the sciatic nerve. Exparel in this situation is being used off-label given that it is not FDA-approved for lower extremity nerve blocks. However, Exparel is commonly used in other nerve blocks and is FDA-approved for blocks such as the interscalene brachial plexus block.
  Arms: Bupivacaine
Drug: Exparel + Bupivacaine — Patients will receive the ERAS standard of care which includes gabapentin, Tylenol, and Toradol or Celebrex preoperatively as well as 20 cc of 0.25% bupivacaine injected in the adductor space followed by 30 cc of 0.25% bupivacaine in the sciatic nerve block. Injections will be completed by an anesthesia provider in the same manner as above. Catheters will be left in both spaces with post-operative pumps running 0.2% ropivacaine at 8 cc/hr.
  Arms: Exparel + Bupivacaine

SUMMARY:
This study will compare the use of single-shot Exparel, a long-acting local anesthestic, with the use of catheters that deliver a continuous flow of the short-acting local anesthetic ropivacaine. The comparison will be done in patients who receive preoperative adductor and sciatic nerve blocks prior to orthopedic surgery for traumatic lower extremity injury. The patients' pain will then be monitored for up to 72 hours after injection, measuring every 12 hours after injection until the 72-hour mark. Opioid consumption (measured in morphine milligram equivalents) will also be tracked over this time period.

DETAILED DESCRIPTION:
The use of Exparel has been widely criticized over the past few years with regard to its efficacy compared to perineural catheters and whether or not it truly lasts 72 hours, as is often advertised. However, it is still used in many centers for the proposed increased duration of action and ease of use compared to indwelling catheters, which require a greater degree of monitoring and follow-up for removal. Various studies conducted have looked at the efficacy of Exparel and have found no superiority over nerve blocks with other local anesthetic agents. However, nerve blocks with catheters have never been directly compared to exparel injections for pain control. As such, the goal of this study is to elucidate whether there truly is a difference between the two. In this study, the study team will compare preoperative adductor and sciatic nerve blocks with exparel versus catheters in orthopedic surgery patients who present with a traumatic lower extremity injury. Exparel has been documented to increase the duration of a nerve block by up to 72 hours. Studies comparing exparel single shot versus bupivacaine single shot have favored for the latter, which pharmacodynamically makes sense. A liposomal compound which slowly denatures to present an active component would seemingly be unlikely to match up against the higher concentration of said active component flood the desired site of action. In our study, the study team plans to measure the duration of the block with the addition of exparel in comparison to the duration of the block with a catheter which is connected to a pump continuously infusing a set rate of local anesthetics. Our primary research question is whether there is a statistically significant difference in pain control for 72 hours post-op in lower extremity orthopedic trauma when using Exparel versus a short-acting local anesthetic supplied via continuous infusion, in this case ropivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Closed lower extremity orthopedic injury
* Opioid naive patients
* No other significant surgical injuries on admission as determined by study physician

Exclusion Criteria:

* Allergy to local anesthetics
* Multiple traumatic injuries
* Weight less than 60 kg
* Prior opioid use or risk of increased pain control needs as determined by PI
* Chronic opioid use
* Open fractures
* Plastic surgery needed for complete closure
* Patient has intraoperative cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2028-08-11 (Estimated); Study Completion 2029-08-11 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score | 12 hours
  Visual Analog Scale on a scale of 0-10 (0 is no pain and 10 is the worst pain)
Postoperative Pain Score | 24 hours
  Visual Analog Scale on a scale of 0-10 (0 is no pain and 10 is the worst pain)
Postoperative Pain Score | 36 hours
  Visual Analog Scale on a scale of 0-10 (0 is no pain and 10 is the worst pain)
Postoperative Pain Score | 48 hours
  Visual Analog Scale on a scale of 0-10 (0 is no pain and 10 is the worst pain)
Postoperative Pain Score | 60 hours
  Visual Analog Scale on a scale of 0-10 (0 is no pain and 10 is the worst pain)
Postoperative Pain Score | 72 hours
  Visual Analog Scale on a scale of 0-10 (0 is no pain and 10 is the worst pain)

SECONDARY OUTCOMES:
Morphine equivalents | Day 1
  Morphine equivalents at 24 hours postoperatively
Morphine equivalents | Day 2
  Morphine equivalents at 24-48 hours postoperatively
Morphine equivalents | Day 3
  Morphine equivalents at 48-72 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- The George Washington University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No